CLINICAL TRIAL: NCT04788680
Title: Assessment of the Effects of Non-calorie Sweeteners on Gut Barrier and Inflammatory Markers Compared to Those of Sugars in Healthy Individuals
Brief Title: Effects of Non-calorie Sweeteners, Mono- and Disaccharides on Intestinal Barrier Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ina Bergheim, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UVienna21
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Dietary Habits; Endotoxemia
MeSH Terms: conditions — Feeding Behavior; Endotoxemia

STUDY DESIGN:
Intervention Model Description: All participants receive all interventional diets
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Beverage 1 (Experimental): Participants receive a beverage with a defined amount of non-nutritive sweetener.
  Interventions: Other: Dietary intervention 1
- Experimental: Beverage 2 (Experimental): Participants receive a beverage with a defined amount of non-nutritive sweetener.
  Interventions: Other: Dietary Intervention 2
- Experimental: Beverage 3 (Experimental): Participants receive a beverage with a defined amount of monosaccharide.
  Interventions: Other: Dietary Intervention 3
- Experimental: Beverage 4 (Experimental): Participants receive a beverage with a defined amount of disaccharide.
  Interventions: Other: Dietary Intervention 4

INTERVENTIONS:
Other: Dietary intervention 1 — Participants receive a beverage with a defined amount of non-nutritive sweetener.
  Arms: Experimental: Beverage 1
Other: Dietary Intervention 2 — Participants receive a beverage with a defined amount of non-nutritive sweetener and maltodextrin.
  Arms: Experimental: Beverage 2
Other: Dietary Intervention 3 — Participants receive a beverage with a defined amount of monosaccharide.
  Arms: Experimental: Beverage 3
Other: Dietary Intervention 4 — Participants receive a beverage with a defined amount of disaccharide.
  Arms: Experimental: Beverage 4

SUMMARY:
The aim of the present study is to determine the effect of non-nutritive sweeteners on intestinal barrier function and inflammatory markers in healthy subjects in comparison to mono- and disaccharides.

DETAILED DESCRIPTION:
In the intervention study normal weight participants will receive beverages sweetened with non-nutritive sweeteners, mono- and disaccharides for a defined number of days. Before and after intervention parameters of intestinal barrier function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* No known history of metabolic diseases/disorders
* BMI <25 kg/m2

Exclusion Criteria:

* Food allergies or intolerances (esp. fructose intolerance and malabsorption)
* Chronic disease of the gastrointestinal tract
* Renal insufficiency
* Taking drugs affecting lipid or glucose metabolism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in parameters of intestinal barrier function. | 1 week
  Changes in plasma endotoxin levels.
Changes in inflammatory markers. | 1 week
  Changes in IL-6 plasma levels (ng/ml).

SECONDARY OUTCOMES:
Changes in blood pressure. | 1 week
  Changes in systolic and diastolic blood pressure
Changes in markers for glucose metabolism. | 1 week
  Changes in fasting glucose (mg/dl) and fasting insulin levels (mU/l)
Changes in markers for glucose metabolism. | 1 week
  Changes in fasting insulin levels (mU/l).
Changes in blood lipid levels. | 1 week
  Changes in triglyceride levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No